CLINICAL TRIAL: NCT00603694
Title: Hippocampal Radiation Exposure and Memory: A Pilot Study
Brief Title: Hippocampal Radiation Exposure and Memory
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 07-0023-CE
Record Dates: First submitted 2008-01-16; First posted 2008-01-29 (Estimated); Last update posted 2016-06-23 (Estimated); Status verified 2016-06

CONDITIONS: Arteriovenous Malformation; Schwannoma; Trigeminal Neuralgia
Keywords: Hippocampus; Memory; Radiation
MeSH Terms: conditions — Arteriovenous Malformations; Neurilemmoma; Trigeminal Neuralgia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- 1: (Experimental group): Receiving > 2 Gy SRS to left hippocampus (n=10)
- 2: (Low-dose control group): Receiving < 0.5 Gy SRS to left hippocampus (n=10)
- 3: (High-dose control group): Receiving whole brain PCI (n=10)

SUMMARY:
Neurocognitive impairment as a result of gamma knife radiosurgery has not been well studied and is poorly understood. Radiosurgery to the base of skull for the treatment of benign and malignant disorders may consequently impair memory function. There is a need to evaluate changes in memory function that may be associated with such exposures.

In this pilot study, we will investigate changes in hippocampal-dependent memory function in 10 patients receiving a low SRS dose to the hippocampus. We will also investigate such changes in a no-dose control group and a high-dose control group. This study will provide preliminary estimates of variance in memory changes associated with radiation exposure, and will then permit us to design future studies with the appropriate sample size justification.

ELIGIBILITY:
Inclusion Criteria:

* Patients planned for radiosurgery for benign disorders (Groups 1&2).
* Patients planned for prophylactic cranial irradiation (Group 3)

Exclusion Criteria:

* Previous cranial radiation
* Severe psychiatric disorder
* Severe cognitive or memory impairment (MMSE < 21)
* Non-English speaking, which will potentially make memory testing difficult and unreliable.
* Other medical conditions deemed by the PI or associates to make the patient ineligible for protocol procedures
* Patients on steroid medications.
* Left hand dominant patients
* Dose exposure to left hippocampus >0.5Gy and <2Gy. We will attempt to estimate dose to hippocampus prior to enrollment using pre-planning on diagnostic imaging to minimize exclusion of patients due to dose exposure >0.5 Gy and < 2Gy following baseline memory testing.
* Benzodiazepine or narcotics given on the day of radiotherapy/radiosurgery prior to completion of the study procedures
* Previous brain surgery within one year prior to radiosurgery
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have consented to GK radiosurgery or cranial radiation.
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2007-09; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Joey & Toby Tanenbaum Gamma Knife Centre, Toronto Western Hospital, Toronto, Ontario, Canada